CLINICAL TRIAL: NCT04905524
Title: Activity Changes in Irritable Bowel Syndrome (IBS), Anxiety, and Depression Following the Use of Viome Precision Nutrition Program (VPNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viome (Industry)
Responsible Party: Principal Investigator, Momchilo Vuyisich, Study Principal Investigator, Viome
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: V216
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Depression, Anxiety; IBS - Irritable Bowel Syndrome
Keywords: Depression; Anxiety; Irritable bowel syndrome; Viome precision nutrition program; VNPN; IBS; PHQ9; GAD7; ROME-IV; Viome; Diet; Nutrition; Supplements
MeSH Terms: conditions — Depression; Anxiety Disorders; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a single group cohort study; the first cohort consists of participants with self reported Irritable Bowel Syndrome (IBS), the second cohort consists of participants with self reported depression and the last cohort consists of participants with self reported anxiety.
  All cohorts receive diet and supplement recommendations from Viome based on participants' sample results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): All participants received the intervention in this trial (VPNP diet and supplement recommendations).
  Interventions: Dietary Supplement: VIOME Precision Nutrition Program

INTERVENTIONS:
Dietary Supplement: VIOME Precision Nutrition Program — Diet and supplements recommendations
  Other Names: VPNP

SUMMARY:
Viome costumers are consented and recruited for this study and complete the questionnaires upon enrollment. Any participant who previously self reported depression, anxiety, or Irritable Bowel Syndrome (IBS) qualify for this study.

All participants receive Viome's diet, supplement and recommendations.

DETAILED DESCRIPTION:
Participants receive Viome Precision Nutrition Program (VPNP) after completing the health assessment and questionnaire. VPNP consists of diet, supplement and recommendations based on results from their sample results and their self reported questionnaire.

After approximately 5 months, participants were given the same health assessment questionnaire.

The results and data collected before and after the VPNP are analyzed to find correlations and differences between the measurements taken at the beginning of the trial and again approximately 5 months after.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 score 5 or above
* GAD-7 score 5 or above
* IBS ROME-IV score 125 or above
* Females and males aged 18 years or older
* Signed and dated informed consent prior to any trial-specific procedures are performed
* Able to speak and read English
* Willing and able to follow the trial instructions
* Viome existing costumer

Exclusion Criteria:

* Unable/unwilling to complete the provided questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Disease activity changes for IBS | ~5 months
  Change of disease activity measurements in participants with self reported IBS after they have received Viome Precision Nutrition Program (VPNP), which consists of dietary supplement recommendations from Viome using clinically validated questionnaires. For IBS, Rome IV classification and criteria based on interpretation and self reporting of IBS, experience and symptoms were used to measure before and after VPNP for approximate duration of 5 months.
Disease activity changes depression | ~5 months
  Change of disease activity measurements in participants with self reported depression after they have received Viome Precision Nutrition Program (VPNP), which consists of dietary supplement recommendations from Viome using clinically validated questionnaires. For depression, brief patient health questionnaire mood scale (PHQ-9) was used.
Disease activity changes anxiety | ~5 months
  Change of disease activity measurements in participants with self reported anxiety after they have received Viome Precision Nutrition Program (VPNP), which consists of dietary supplement recommendations from Viome using clinically validated questionnaires. For anxiety, General Anxiety Disorder 7 (GAD-7) was used, which is designed to assess the participants' health status during the previous 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Momo Vuyisich, PhD, Principal Investigator — Viome
Locations (1):
- Viome Research Institute, Bothell, Washington, United States

IPD SHARING:
Plan to Share IPD: No